CLINICAL TRIAL: NCT03762486
Title: The Effects of Two Different Electrical Stimulation Methods on the Pain Intensity of the Patients Who Had Undergone Abdominal Surgery With a Midline Incision: Randomized Controlled Clinical Trial
Brief Title: The Pain Intensity of the Patients Who Had Undergone Abdominal Surgery With a Midline Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Bediye Oztas, Teaching Staff, Yuksek Ihtisas University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: YuksekIU
Record Dates: First submitted 2018-01-05; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-03

CONDITIONS: Transcutaneous Electric Nerve Stimulation
Keywords: Postoperative pain; Alternative therapy; Acupuncture; TENS; Surgical nursing; Randomised controlled trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: TENS was applied to around the insicion: Transcutaneous electrical nerve stimulation was applied to around the incision.
  TAES was applied to acupuncture points: Transcutaneous electrical stimulation was applied to acupuncture points.
  No intervention: No stimulation was performed to the patients.
  A standard analgesia protocol for post-operative pain control was used in all patients included in the study. A standard antiemetic protocol was used for all patients after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS to around the incision (Active Comparator): The Patient Controlled Analgesia infusion was started right after the surgery. TENS was applied to around the incision.
  Interventions: Other: TENS
- TAES to the acupuncture points (Active Comparator): The Patient Controlled Analgesia infusion was started right after the surgery. TAES was applied to acupuncture points.
  Interventions: Other: TAES
- No stimulation (No Intervention): No stimulation was performed to the patients in the control group.

INTERVENTIONS:
Other: TENS — 4 electrodes were placed 2-3 cm lateral to the incision of the patients at the 30th minute and 2, 18, 22, 42, and 46th hours after the surgery and electrical stimulation was implemented at varying frequencies of 2-100 Hz for 30 minutes, at a maximum current intensity of 12 milliamperes that would not bother the patient or create muscle contractions, with a pulse duration of 0.25 min
  Other Names: First Intervention Group
  Arms: TENS to around the incision
Other: TAES — 4 electrodes were placed at the ST25, P6, ST36, and LI4 acupuncture points of the patients at the 30th minute and 2, 18, 22, 42, and 46th hours after the surgery and electrical stimulation was implemented at varying frequencies of 2-100 Hz for 30 minutes, at a maximum current intensity of 12 milliamperes that would not bother the patient or create muscle contractions, with a pulse duration of 0.25 min
  Other Names: Second Intervention Group
  Arms: TAES to the acupuncture points

SUMMARY:
The purpose of this study is to determine the effects of transcutaneous electrical nerve stimulation (TENS) and transcutaneous acupoint electrical stimulation (TAES) on pain and analgesic drug consumption in patients who had undergone abdominal surgery with a midline incision. Evidence for the effects of and transcutaneous electrical stimulation on pain and analgesic consumption on patients undergoing abdominal surgery with severe pain experience and high levels of neuroendocrine stress response is uncertain.

DETAILED DESCRIPTION:
This research was conducted as a randomized controlled trial. 158 patients who had undergone abdominal surgery with diagnosis of gastric and colorectal cancer were assessed for eligibility. This research sample consisted of 48 patients who underwent abdominal surgery with a midline incision. The patients were randomized into three groups, the first intervention group, which used TENS (around the incision), the second intervention group, which used TAES (ST25, P6, ST36, Lİ4 acupuncture points) and the control group, which did not. Electric stimulation was performed at the 30th minute, second, 18th, 21st, 40th, and 45th hours after the operation. Pain scores and analgesic consumption were assessed in the first 48 hours after surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an American Society of Anesthesiologists (ASA) score of I-II
* Patients were aged over 18 years
* Patients who could read and write Turkish
* Patients who were scheduled to undergo elective abdominal surgery with a midline incision for a diagnosis of stomach or colorectal cancer
* Patients without any impairment of vision, hearing or speech

Exclusion Criteria:

* Patients who had a pacemaker
* Patients whose skin integrity around the incision was degraded
* Patients had a cognitive disorder, had a history of chronic pain, or were suffering from neurological, renal, cardiac or pulmonary disorders that could affect the test results
* Patients with an opioid addiction
* Patients those who had previously undergone electrical stimulation treatment
* Morbidly obese subjects
* Patients using psychoactive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | The pain levels were evaluated and compared within postoperative first 48 hours.
  First Intervention Group: Electrical stimulation was implemented at the 30th minute and 2, 18, 22, 42, and 46th hours after the surgery.
  Second Intervention Group: Electrical stimulation was implemented at acupuncture points of the patients at the 30th minute and 2, 18, 22, 42, and 46th hours after the surgery.
  Control Group: No intervention was performed to the patients in the control group.
  The pain intensity of each groups' patients were recorded and compred at the post-operative 2, 18, 22, 42, and 46th hours. Pain intensity was evaluated with VAS. VAS with a range of 1-10 points was used while evaluating the pain intensity of all patients .The increase of the scale score shows that the pain intensity increases.

SECONDARY OUTCOMES:
Nausea severity | The nausea severity of the patients were evaluated at the periods of 0-6, 6-24, 24-48 hours. Patients were assessed in postoperative first 48 hours.
  VAS with a range of 1-10 points was used while evaluating the nausea severity of all patients .The increase of the scale score shows that the nausea severity increases.
Antiemetic drug consumption | Antiemetic drug consumption of the patients was evaluated at the periods of 0-24 and 24-48 hours. Patients were assessed in postoperative first 48 hours.
  The antiemetic drug amount administered to the patients was recorded in mg.
Pulmonary function tests | Pulmonary function evaluations of the patients were performed at the 24th and 48th hours. Patients were assessed in postoperative first 48 hours.
  The pulmonary functions of the patients were evaluated with a portable spirometer. Peak expiratory flow (PEF) and forced vital capacity (FVC) values were recorded. The measurement of respiratory functions was performed with the patient wrapping the disposable mouthpiece well with the lips during the measurement. The patient was asked to breathe deeply and exhale suddenly and quickly. This process was repeated three times and the best performance was taken as the base value.
Vomiting | Vomiting status of the patients were evaluated at the periods of 0-6, 6-24, 24-48 hours. Patients were assessed in postoperative first 48 hours.
  Vomiting: The number of times the patients vomited was recorded
Analgesic drug consumption | Analgesic drug consumption of the patients was evaluated at the periods of 0-24 and 24-48 hours. Patients were assessed in postoperative first 48 hours.
  All patients were administered intravenous tramadol hydrochloride infusion with the Patient Controlled Analgesia for the first 48 hours. Dexketoprofen trometamol vial intravenous and/or 50 mg. Pethidine hydrochloride intramuscular was used as the rescue analgesic.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Iyigun, Professor, Study Director — Turkish Nurses Society

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breit R, Van der Wall H. Transcutaneous electrical nerve stimulation for postoperative pain relief after total knee arthroplasty. J Arthroplasty. 2004 Jan;19(1):45-8. doi: 10.1016/s0883-5403(03)00458-3. PMID 14716650
- [Background] Wu MS, Chen KH, Chen IF, Huang SK, Tzeng PC, Yeh ML, Lee FP, Lin JG, Chen C. The Efficacy of Acupuncture in Post-Operative Pain Management: A Systematic Review and Meta-Analysis. PLoS One. 2016 Mar 9;11(3):e0150367. doi: 10.1371/journal.pone.0150367. eCollection 2016. PMID 26959661
- [Result] Dias M, Carneiro NM, Guerra LA, Velarde GC, de Souza PA, da Silva LL, de Abreu e Souza RR, Nolasco R, Olej B. Effects of electroacupuncture on local anaesthesia for inguinal hernia repair: a randomised placebo-controlled trial. Acupunct Med. 2010 Jun;28(2):65-70. doi: 10.1136/aim.2009.000570. PMID 20615859
- [Result] Bjersa K, Andersson T. High frequency TENS as a complement for pain relief in postoperative transition from epidural to general analgesia after pancreatic resection. Complement Ther Clin Pract. 2014 Feb;20(1):5-10. doi: 10.1016/j.ctcp.2013.11.004. Epub 2013 Nov 20. PMID 24439637
- [Result] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Result] Chen L, Tang J, White PF, Sloninsky A, Wender RH, Naruse R, Kariger R. The effect of location of transcutaneous electrical nerve stimulation on postoperative opioid analgesic requirement: acupoint versus nonacupoint stimulation. Anesth Analg. 1998 Nov;87(5):1129-34. PMID 9806695
- [Result] Chen Y, Yang Y, Yao Y, Dai D, Qian B, Liu P. Does transcutaneous electric acupoint stimulation improve the quality of recovery after thyroidectomy? A prospective randomized controlled trial. Int J Clin Exp Med. 2015 Aug 15;8(8):13622-7. eCollection 2015. PMID 26550304
- [Result] da Silva MP, Liebano RE, Rodrigues VA, Abla LE, Ferreira LM. Transcutaneous electrical nerve stimulation for pain relief after liposuction: a randomized controlled trial. Aesthetic Plast Surg. 2015 Apr;39(2):262-9. doi: 10.1007/s00266-015-0451-6. Epub 2015 Feb 10. PMID 25665520
- [Result] DeSantana JM, Santana-Filho VJ, Guerra DR, Sluka KA, Gurgel RQ, da Silva WM Jr. Hypoalgesic effect of the transcutaneous electrical nerve stimulation following inguinal herniorrhaphy: a randomized, controlled trial. J Pain. 2008 Jul;9(7):623-9. doi: 10.1016/j.jpain.2008.01.337. Epub 2008 Apr 3. PMID 18387854
- [Result] Engen DJ, Carns PE, Allen MS, Bauer BA, Loehrer LL, Cha SS, Chartrand CM, Eggler EJ, Cutshall SM, Wahner-Roedler DL. Evaluating efficacy and feasibility of transcutaneous electrical nerve stimulation for postoperative pain after video-assisted thoracoscopic surgery: A randomized pilot trial. Complement Ther Clin Pract. 2016 May;23:141-8. doi: 10.1016/j.ctcp.2015.04.002. Epub 2015 Apr 20. PMID 25935320
- [Result] Lan F, Ma YH, Xue JX, Wang TL, Ma DQ. Transcutaneous electrical nerve stimulation on acupoints reduces fentanyl requirement for postoperative pain relief after total hip arthroplasty in elderly patients. Minerva Anestesiol. 2012 Aug;78(8):887-95. Epub 2012 Apr 24. PMID 22531569
- [Result] Feng X, Ye T, Wang Z, Chen X, Cong W, Chen Y, Chen P, Chen C, Shi B, Xie W. Transcutaneous acupoint electrical stimulation pain management after surgical abortion: A cohort study. Int J Surg. 2016 Jun;30:104-8. doi: 10.1016/j.ijsu.2016.04.042. Epub 2016 Apr 29. PMID 27142864
- [Result] Wang H, Xie Y, Zhang Q, Xu N, Zhong H, Dong H, Liu L, Jiang T, Wang Q, Xiong L. Transcutaneous electric acupoint stimulation reduces intra-operative remifentanil consumption and alleviates postoperative side-effects in patients undergoing sinusotomy: a prospective, randomized, placebo-controlled trial. Br J Anaesth. 2014 Jun;112(6):1075-82. doi: 10.1093/bja/aeu001. Epub 2014 Feb 26. PMID 24576720
- [Result] Hong SJ, Lee E. Effect of evidence-based postoperative pain guidelines via web for patients undergoing abdominal surgery in South Korea. Asian Nurs Res (Korean Soc Nurs Sci). 2014 Jun;8(2):135-42. doi: 10.1016/j.anr.2014.05.005. Epub 2014 May 21. PMID 25030646
- [Result] Kara B, Baskurt F, Acar S, Karadibak D, Ciftci L, Erbayraktar S, Gokmen AN. The effect of TENS on pain, function, depression, and analgesic consumption in the early postoperative period with spinal surgery patients. Turk Neurosurg. 2011;21(4):618-24. PMID 22194125
- [Result] Senol Karatas S, Eti Z, Saracoglu KT, Gogus FY. Does perioperative opioid infusion increase postoperative opioid requirement? Agri. 2015;27(1):47-53. doi: 10.5505/agri.2015.71676. PMID 25867874
- [Result] Kayman-Kose S, Arioz DT, Toktas H, Koken G, Kanat-Pektas M, Kose M, Yilmazer M. Transcutaneous electrical nerve stimulation (TENS) for pain control after vaginal delivery and cesarean section. J Matern Fetal Neonatal Med. 2014 Oct;27(15):1572-5. doi: 10.3109/14767058.2013.870549. Epub 2014 Jan 8. PMID 24283391
- [Result] Kehlet H. Procedure-specific postoperative pain management. Anesthesiol Clin North Am. 2005 Mar;23(1):203-10. doi: 10.1016/j.atc.2004.11.001. PMID 15763419
- [Result] Kerai S, Saxena KN, Taneja B, Sehrawat L. Role of transcutaneous electrical nerve stimulation in post-operative analgesia. Indian J Anaesth. 2014 Jul;58(4):388-93. doi: 10.4103/0019-5049.138966. PMID 25197104
- [Result] Hamza MA, White PF, Ahmed HE, Ghoname EA. Effect of the frequency of transcutaneous electrical nerve stimulation on the postoperative opioid analgesic requirement and recovery profile. Anesthesiology. 1999 Nov;91(5):1232-8. doi: 10.1097/00000542-199911000-00012. PMID 10551571
- [Result] Rakel B, Frantz R. Effectiveness of transcutaneous electrical nerve stimulation on postoperative pain with movement. J Pain. 2003 Oct;4(8):455-64. doi: 10.1067/s1526-5900(03)00780-6. PMID 14622666
- [Result] Francis RP, Johnson MI. The characteristics of acupuncture-like transcutaneous electrical nerve stimulation (acupuncture-like TENS): a literature review. Acupunct Electrother Res. 2011;36(3-4):231-58. doi: 10.3727/036012911803634139. PMID 22443026
- [Result] Robleda G, Roche-Campo F, Sanchez V, Gich I, Banos JE. Postoperative Discomfort After Abdominal Surgery: An Observational Study. J Perianesth Nurs. 2015 Aug;30(4):272-9. doi: 10.1016/j.jopan.2014.06.005. Epub 2015 May 16. PMID 26210558
- [Result] Rosen HI, Bergh IH, Oden A, Martensson LB. Patients experiences of pain following day surgery - at 48 hours, seven days and three months. Open Nurs J. 2011;5:52-9. doi: 10.2174/1874434601105010052. Epub 2011 Jul 6. PMID 21769308
- [Result] Sbruzzi G, Silveira SA, Silva DV, Coronel CC, Plentz RD. Transcutaneous electrical nerve stimulation after thoracic surgery: systematic review and meta-analysis of 11 randomized trials. Rev Bras Cir Cardiovasc. 2012 Jan-Mar;27(1):75-87. doi: 10.5935/1678-9741.20120012. English, Portuguese. PMID 22729304
- [Result] Silva MB, de Melo PR, de Oliveira NM, Crema E, Fernandes LF. Analgesic effect of transcutaneous electrical nerve stimulation after laparoscopic cholecystectomy. Am J Phys Med Rehabil. 2012 Aug;91(8):652-7. doi: 10.1097/PHM.0b013e318246638f. PMID 22311059
- [Result] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Result] Gavronsky S, Koeniger-Donohue R, Steller J, Hawkins JW. Postoperative pain: acupuncture versus percutaneous electrical nerve stimulation. Pain Manag Nurs. 2012 Sep;13(3):150-6. doi: 10.1016/j.pmn.2009.08.001. Epub 2010 Jan 6. PMID 22929602
- [Result] Tokuda M, Tabira K, Masuda T, Nishiwada T, Shomoto K. Effect of modulated-frequency and modulated-intensity transcutaneous electrical nerve stimulation after abdominal surgery: a randomized controlled trial. Clin J Pain. 2014 Jul;30(7):565-70. doi: 10.1097/AJP.0b013e31829ea151. PMID 24901753
- [Result] Unterrainer AF, Friedrich C, Krenn MH, Piotrowski WP, Golaszewski SM, Hitzl W. Postoperative and preincisional electrical nerve stimulation TENS reduce postoperative opioid requirement after major spinal surgery. J Neurosurg Anesthesiol. 2010 Jan;22(1):1-5. doi: 10.1097/ANA.0b013e3181b7fef5. PMID 19779370
- [Result] Wang B, Tang J, White PF, Naruse R, Sloninsky A, Kariger R, Gold J, Wender RH. Effect of the intensity of transcutaneous acupoint electrical stimulation on the postoperative analgesic requirement. Anesth Analg. 1997 Aug;85(2):406-13. doi: 10.1097/00000539-199708000-00029. PMID 9249122
- [Result] Ward CW. Procedure-specific postoperative pain management. Medsurg Nurs. 2014 Mar-Apr;23(2):107-10. PMID 24933788
- [Result] Yeh ML, Chung YC, Chen KM, Tsou MY, Chen HH. Acupoint electrical stimulation reduces acute postoperative pain in surgical patients with patient-controlled analgesia: a randomized controlled study. Altern Ther Health Med. 2010 Nov-Dec;16(6):10-8. PMID 21280458
- [Result] Yeh ML, Chung YC, Chen KM, Chen HH. Pain reduction of acupoint electrical stimulation for patients with spinal surgery: a placebo-controlled study. Int J Nurs Stud. 2011 Jun;48(6):703-9. doi: 10.1016/j.ijnurstu.2010.10.009. Epub 2010 Nov 30. PMID 21122849
- See also: for access to resources — https://www.ncbi.nlm.nih.gov/pubmed/citmatch
- Available data/document: Individual Participant Data Set — https://www.ncbi.nlm.nih.gov/pubmed/citmatch

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03762486/Prot_SAP_000.pdf